CLINICAL TRIAL: NCT03077633
Title: Cervical Cerclage for Twin Pregnancy With Sonographic Cervical Length 0.1 to 15.0 mm: A Randomized Clinical Trial
Brief Title: Cerclage for Twins With Short Cervix
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Financial/business decision by Sponsor to not proceed with this study
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OBX0038
Record Dates: First submitted 2017-03-03; First posted 2017-03-13 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Preterm Birth; Preterm Labor With Preterm Delivery, Unspecified Trimester, Fetus 2; Cervical Incompetence; Cervical Shortening
Keywords: Cerclage; Cervical shortening; Twins; Progesterone
MeSH Terms: conditions — Premature Birth; Uterine Cervical Incompetence | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Two groups: Cerclage + Progesterone vs. Progesterone alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cervical Cerclage + Progesterone (Active Comparator): Placement of a Cervical Cerclage plus the daily administration of vaginal progesterone (200mg tab)
  Interventions: Procedure: Cervical Cerclage placement; Drug: Vaginal Progesterone
- Progesterone (Placebo Comparator): Daily administration of vaginal progesterone (200mg tab)
  Interventions: Drug: Vaginal Progesterone

INTERVENTIONS:
Procedure: Cervical Cerclage placement — Cervical Cerclage placement
  Arms: Cervical Cerclage + Progesterone
Drug: Vaginal Progesterone — 200mg tab of vaginal progesterone administered daily from time of randomization until delivery.
  Other Names: Prometrium

SUMMARY:
A prospective randomized control trial that will compare cervical cerclage plus vaginal progesterone to vaginal progesterone along in twin pregnancies complicate by a short cervix (</= 15.0mm) between 16w0d to 25w6d.

DETAILED DESCRIPTION:
A prospective Randomized Trial that will test whether treatment with cervical cerclage plus vaginal progesterone improves pregnancy outcomes among women with twin pregnancy at 16 0/7 to 25 6/7 weeks of gestation who have a cervical length (CL) of 0.1 to 15.0 mm on transvaginal ultrasound exam, the rate of preterm birth at less than 32 weeks of gestation (PTB<32 wks.) and the rate of adverse perinatal outcome will be lower in those treated with cervical cerclage plus vaginal progesterone than in those treated with vaginal progesterone alone.

ELIGIBILITY:
Inclusion Criteria:

* Twin pregnancy (see Exclusion Criterion (a) below re: monochorionic twins)
* Gestational age 16 0/7 to 25 6/7 weeks at time of enrollment by best-estimated age.
* Cervical length 0.1 to 15.0 mm on transvaginal ultrasound examination. (Cervical length is taken to mean the length of the closed portion of the cervical canal.

Exclusion Criteria:

* Maternal age less than 18 years
* Monochorionic twins (such as monochorionic-diamniotic, monochorionic-monoamniotic, or conjoined twins)
* Rupture of membranes, either twin
* One or both twins has no cardiac activity
* One or both twins has known or suspected major malformation, aneuploidy, or polyhydramnios
* Maternal congenital uterine anomaly (such as bicornuate uterus, unicornuate uterus)
* Pregnancy started as triplets or higher-order multifetal gestation and then reduced to twins, either spontaneously or via procedure
* Symptomatic uterine contractions, 6 or more per hour
* Ongoing bleeding from uterus
* Patient declines to consider cerclage
* Patient declines treatment with vaginal progesterone
* Allergy to progesterone or peanuts (because the vaginal progesterone formulation used will be a capsule of micronized progesterone in peanut oil.)
* Cerclage is already in place
* Cerclage placement is judged to be technically impossible
* Patient has a history of poor follow-up or poor adherence to physician recommendations
* Patient is planning to relocate outside the local area before the end of pregnancy such that delivery records will be unavailable
* Patient does not give consent to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Rate of very preterm birth (PTB) | Time frame measured on the date the infant is born. We anticipate this time frame to be approximately 16 weeks.
  Rate of very PTB (PTB less than 32 weeks)
Rate of adverse perinatal outcome | Time frame measured 28 days after the infant is born. We anticipate this time frame to be approximately 28 weeks.
  The rate of adverse perinatal outcome defined as any one or more of the following: Miscarriage, stillbirth, neonatal death, respiratory distress syndrome, bronchopulmonary dysplasia, intraventricular hemorrhage (grade III or IV), necrotizing enterocolitis, culture proven sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Combs, MD, Principal Investigator — Pediatrix

IPD SHARING:
Plan to Share IPD: Undecided